CLINICAL TRIAL: NCT01839006
Title: Clinical Significance of Supranormal Differential Renal Function in the Recovery of Unilateral Hydronephrosis After Surgery: Long-term Results
Brief Title: Clinical Significance of Supranormal Differential Renal Function in the Recovery of Hydronephrosis
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Cho, Seoul National University Hospital, Seoul National University Hospital
Other Study IDs: supranormal; supranormal DRF
Record Dates: First submitted 2011-06-25; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Hydronephrosis
Keywords: hydronephrosis; ultrasonography; Kidney Function Test; Patients with unilateral UPJO and patients with preop HN in USG and supranormal renal function in DTPA renography
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with supranormal renal function: Patients with preoperative HN and supranormal renal function in DTPA renography
  Interventions: Procedure: dismembered pyeloplasty

INTERVENTIONS:
Procedure: dismembered pyeloplasty — Using a flank approach, as the patient was placed in the lateral decubitus position, and an anterior subcostal incision was made. The narrow segment of UPJ was identified and resected, and then the proximal edge of the ureter was spatulated to allow a wide anastomosis between the ureter and the most dependent part of the renal pelvis. The extent of renal pelvis reduction was decided by the surgeon.

SUMMARY:
The purpose of this study is to assess the clinical significance of supranormal differential renal function (DRF) in the recovery of unilateral hydronephrosis (HN) after surgery, pediatric patients who underwent pyeloplasty for ureteropelvic junction obstruction (UPJO) who showed supranormal DRF (> 55%) in the DTPA renography will be analyzed.

DETAILED DESCRIPTION:
To assess the clinical significance of supranormal differential renal function (DRF) in the recovery of unilateral hydronephrosis (HN) after surgery, pediatric patients who underwent pyeloplasty for ureteropelvic junction obstruction (UPJO) who showed supranormal DRF (> 55%) in the DTPA renography will be analyzed. Clinical parameters including age at the first visit, age at operation, gender, laterality, and follow-up period will be evaluated. To evaluate predictors of recovery from supranormal renal function according to the level of DRF, univariate and multivariate logistic regression analyses will be performed. Patients would be subcategorized into two groups; group A (DRF ≤60%) and group B (DRF >60%) in consideration of the mean value of preoperative DRF and each parameter of group A was compared to that of group B using independent sample's t test and chi square test. Kaplan-Meier analysis and log-rank test will be used to determine the difference of recovery time of obstructed hydronephrosis in each parameter.

ELIGIBILITY:
Inclusion Criteria:

* ureteropelvic junction obstruction
* hydronephrosis
* differential renal function more than 55% in DTPA
* follow-up period more than 1 year

Exclusion Criteria:

* urological anomalies, such as vesicoureteral reflux, ureterocele, cystic kidney disease, posterior urethral valves, duplex anomalies, neurogenic bladder, and solitary kidney or patients who underwent any previous urological surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with unilateral UPJO pediatric patients who underwent dismembered pyeloplasty and preoperative HN in USG and supranormal renal function in DTPA renography
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hydronephrosis | postop 6 months
  The grade of hydronephrosis would be check at 6 months postoperatively.

SECONDARY OUTCOMES:
renal parenchymal thickness | postop 6 months
  Renal parenchymal thickness was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, M.D., Principal Investigator — Seoul National Universitiy Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea